CLINICAL TRIAL: NCT02793180
Title: Gulf Documentation of Ambulatory Sick Patients With Heart Failure Registry
Brief Title: Documentation of Heart Failure in a Gulf Registry
Acronym: DYSPNEA
Status: Completed | Type: Observational
Sponsor: Gulf Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: CLCZ696BKW01T
Record Dates: First submitted 2016-05-15; First posted 2016-06-08 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
In the Middle East and the Gulf, the general population have high cardiovascular risks like diabetes, hypertension, smoking and obesity. The average age of a patient with an acute coronary syndrome (ACS) event is relatively young compared to Western populations. Women are multiparous and the rates of consanguinity marriages are high in this region of the world. These risk factors and conditions result in heart failure. Great deal of knowledge is missing regarding the influence of these risk factors on heart failure presentation, the causes and management of heart failure in ambulatory patients in this region of the world.

ELIGIBILITY:
Inclusion Criteria:

1. Is over the age of 21.
2. Has been diagnosed with heart failure, regardless of cause.
3. Is presenting to the outpatient clinic of an internist or cardiologist for follow up.
4. Provides a written consent.

Exclusion Criteria:

1. Prior enrolment in this study.
2. Refusal or inability to provide consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4,000 patients already diagnosed with heart failure. Expected number of patients from each country: Kuwait 1200, Oman 1200, UAE 600, Bahrain 600 and Qatar 400.
Sampling Method: Probability Sample
Enrollment: 3680 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Quantifying the causes of heart failure in the ambulatory patients in the outpatient setting | Single time point at baseline upon inclusion (cross-sectional)
  Number of participants with main reason due to heart failure from Coronary Artery Disease (CAD), Hypertension, Valvular, Idiopathic Dilated Cardiomyopathy, Congenital, Pregnancy / delivery related, or other reason to be specified

SECONDARY OUTCOMES:
Measure investigations that heart failure patients undergo | Up to 6 months before inclusion
  Number of participants who have had echocardiography done less than 1 month, 1-6 months, greater than 6 months from enrollment
Measuring patient functional status in heart failure patients | Single time point at baseline upon inclusion (cross-sectional)
  * Number of participants who can walk independently, walk with assistance, or are unable to walk.
  * Number of participants who are limited in dressing, somewhat limited, or not limited.
  * Number of participants who are can shower in a limited manner, somewhat limited, or not limited
Relationship between cardiovascular risk factors and heart failure | Single time point at baseline upon inclusion (cross-sectional)
Measuring Management Gaps in heart failure patients | Past 12 months upon inclusion
  * Number of participants with 0, 1, 2, or greater than 2 emergency room visits related to heart failure
  * Number of participants with 0,1, 2, or greater than 2 hospital admissions related to heart failure

OTHER OUTCOMES:
Quantifying the distribution of heart failure types | Single time point at baseline upon inclusion (cross-sectional)
  Number of participants that will either have preserved or reduced left ventricular systolic function

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Zubaid, Principal Investigator — Gulf Heart Association
Locations (5):
- Kuwait (5):
  - Adan Hospital, Kuwait City
  - Amiri Hospital, Kuwait City
  - Chest Hospital, Kuwait City
  - Farwanya Hospital, Kuwait City
  - Mubarak Al Kabeer, Kuwait City

REFERENCES:
- [Derived] Zubaid M, Rashed W, Ridha M, Al-Jarallah M, Hamad A, Al Banna R, Sulaiman K, Bazargani N, Almahmeed W, Al Mulla A, Baslaib F, Asaad N, Attur S. Design and Rationale of Gulf Documentation of Ambulatory Sick Patients with Heart Failure (Gulf DYSPNEA) Registry. Heart Views. 2018 Jul-Sep;19(3):81-84. doi: 10.4103/HEARTVIEWS.HEARTVIEWS_9_18. PMID 31007855